CLINICAL TRIAL: NCT04965207
Title: EvaLuAtion On the cHaracteristics of the True/False lUmen and Its Prognostic Value for cOronary CTO Patients Just Before Stent Implantation (LAOHUOJI): a CTO All-comer Register Study
Brief Title: EvaLuAtion On the cHaracteristics of the True/False lUmen and Its Prognostic Value for cOronary CTO Patients Just Before Stent Implantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief physician, Shanghai 10th People's Hospital
Other Study IDs: LAOHUOJI
Record Dates: First submitted 2021-07-11; First posted 2021-07-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion; Intravascular Ultrasound; Percutaneous Coronary Intervention; True Lumen; False Lumen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IVUS will be used to evaluate the ratio of false lumen to occluded segment, the ratio of false lumen to stent length, the location characteristics of false lumen and its prognostic value for perioperative complications, 1-year late lumen loss and MACCE events in patients with coronary CTO.

DETAILED DESCRIPTION:
At present, novel technologies of CTO interventional therapy become mature. These technologies usually artificially cause dissection of coronary artery. The events such as collateral vessel loss, vascular injury and tear, perforation, pericardial tamponade caused by false lumen may theoretically affect the perioperative and long-term prognosis of patients. In this study, intravascular ultrasound (IVUS) was used to evaluate the characteristics of true lumen and false lumen in CTO segment, so as to determine its impact on the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old;
* be diagnosed with CTO;
* CTO located in an epicardial coronary artery with a reference diameter of ≥ 2.5mm;
* comply with all the evaluations and follow-up protocols.

Exclusion Criteria:

* suffered from acute myocardial infarction within the previous 3 months;
* rheumatic valvular disease;
* severe arrhythmia;
* lesions unsuitable for PCI;
* severely abnormal hematopoietic systems, such as platelet counts <100*10^9/L or > 700*10^9/L and white blood cell counts < 3*10^9/L;
* with active bleeding or bleeding tendencies(active ulcers, short-term ischemic stroke, history of hemorrhagic stroke, intracranial space occupying lesions, recent craniocerebral trauma, and other bleeding or bleeding tendency);
* severe coexisting conditions, including severe renal function dysfunction [Glomerular filtration rate less than 60ml/min • 1.73 m2), severe hepatic dysfunction [glutamic-pyruvic transaminase (ALT) or glutamic-oxal acetic transaminase (ALT) elevated more than three times that of the upper limit of the normal reference], severe heart failure (NYHA classification III-IV), acute infectious diseases and immune disorders; tumors; surgery within 3 months;
* a life expectancy less than 12 months;
* pregnancy or planning to become pregnant;
* history of allergy or adverse reactions to aspirin, clopidogrel, ticagrelor, stains, contrast material, anticoagulant, or stents;
* cannot tolerate dual antiplatelet treatment;
* unable to communicate due to cognitive impairment, auditory, or visual impairment;
* participating in another trial for medication or an apparatus and in which the main endpoint has not been reached, or plan to participate in a clinical trial within 12 months of the intervention.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CTO PCI at each of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss | 1 year after PCI
  Late Lumen Loss was defined as the difference between post-stenting minimal lumen diameter (MLD) minus MLD at the time of follow-up.

SECONDARY OUTCOMES:
Late Lumen Loss | 3 year after PCI
  Late Lumen Loss was defined as the difference between post-stenting minimal lumen diameter (MLD) minus MLD at the time of follow-up.
Major Adverse of Cardiovascular and Cerebrovascular Events(MACCE) | Within the first week after PCI, at the 1-year follow-up and at the 3-year follow-up
  including any of the following adverse events before hospital discharge: death from any cause, Q-wave myocardial infarction, recurrent symptoms Heart and Vessels requiring urgent repeat target vessel revascularization with PCI or CABG, tamponade requiring either pericardiocentesis or surgery, and stroke.
Complications | Within the first week after PCI
  Any periprocedural complication was defined as the composite of death, myocardial infarction, stent thrombosis, stroke, vessel perforation, vascular access complications, need for emergency surgical intervention or PCI, and hemoglobin reduction by >3 g/dL.

IPD SHARING:
Plan to Share IPD: Undecided